CLINICAL TRIAL: NCT04292990
Title: A Comparison of Oral Controlled-release Morphine With Transdermal Fentanyl in Nasopharyngeal Cancer Patients With Moderate or Severe Oral Mucositis Pain Induced by Chemoradiotherapy
Brief Title: Comparison of Transdermal Fentanyl and Morphine for Oral Mucositis Pain in Nasopharyngeal Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiarong Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Jiarong Chen, MD, Principal Investigator, Jiangmen Central Hospital
Organization: Jiangmen Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JM0019001
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Pain; Nasopharyngeal Carcinoma; Head and Neck Cancer; Radiation Induced Oral Mucositis
MeSH Terms: conditions — Pain; Nasopharyngeal Carcinoma; Head and Neck Neoplasms | interventions — Fentanyl; Morphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl (Experimental): Intervention: Drug: Fentanyl Transdermal Patch
  Interventions: Drug: Fentanyl
- Morphine (Active Comparator): Intervention: Drug: Morphine Controlled-Release Tablets
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl — Patch releasing drug at the rate of 25 µg/hour, increasing by 25 µg/hour increments to maintain the NRS score≤3 after the frst 24 hours according to no change in pain control. The maximum dose allowed in this study is 300 µg/hour.
  Other Names: Duragesic
  Arms: Fentanyl
Drug: Morphine — Tablets taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. Titration phase: starting at 30 mg, increasing at a minimum of 3 days intervals by 20 mg, with a maximum dose of 100 mg. Maintenance phase: continuing on dose level established in titration phase.
  Other Names: MeiShi KangDing
  Arms: Morphine

SUMMARY:
The primary purpose of this study is to explore the significance of analgesic treatment for radiation-induced oral mucositis pain in patients with nasopharyngeal carcinoma during radiotherapy, and to compare the analgesic effect of morphine controlled-release tablets with that of fentanyl transdermal patch. Half of participants will receive morphine controlled-release tablets,while the other half will receive fentanyl transdermal patch.

DETAILED DESCRIPTION:
Morphine controlled-release tablets and fentanyl transdermal patch each relieve radiation-induced oral mucositis pain in patients with nasopharyngeal carcinoma. But they do so by different mechanisms and in different effects.

Morphine is a classic strong analgesic, which has been widely used in patients with advanced cancer pain. It has achieved satisfactory results in pain control, sleep improvement and quality of life. Oral morphine has been regarded as the standard treatment for moderate and severe cancer pain.

Fentanyl transdermal patch is a system device for transdermal delivery of drugs. It is compressed on a film containing fentanyl memory. The film can continuously release fentanyl into the blood circulation and maintain stable for more than 72 hours. It is not affected by gastrointestinal PH or food, and it has no hepatic frst-pass effect, with a bioavailability of up to 92%.

This study will test the efficacy and safety of morphine controlled-release tablets compared to fentanyl transdermal patch in the treatment of pain in patients with radiation-induced oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Patients were pathologically newly diagnosed with nasopharyngeal carcinoma and had no previous history of other tumors
* According to the treatment strategies of doctors, patients need to receive radiotherapy with or without chemotherapy (for example, neoadjuvant chemotherapy, concurrent chemotherapy, adjuvant chemotherapy) or targeted therapy
* Never use a opioid before treatment
* Hematology: WBC≥4.0×109/L, ANC≥1.5×109/L, PLT≥100×109/L,Hb≥90g/L.
* Participants with the ability to assess the pain level
* Willingness to return to enrolling institution for follow-up

Exclusion Criteria:

* Patients do not conform to the inclusion criteria
* Known allergy to fentanyl, morphine, or any known component of the drug formulation
* Refuse to use of opioid drugs
* Nasopharyngeal patients with mental illness
* Current untreated or unresolved oral candidiasis or oral HSV infection
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Pregnant or Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other contraindications or unsuitable conditions for radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measure | Through chemoradiotherapy completion, 3 weeks
  Self reported pain intensity once a day according to the numeric rating scale (NRS), with 0-10(0=no pain, 10=pain as bad as can be). The higher scores indicate worse pain.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Through chemoradiotherapy completion, 3 weeks
  All adverse events were recorded during treatment, and the skin was examined for local reactions during treatment and after removal of fentanyl transdermal patch.
Quality-of-Life composite Index | Through chemoradiotherapy completion, an average of 2 weeks
  Quality-of-Life was assessed using Karnofsky performance status (KPS) standards of the Union for International Cancer Control and SPAASMS (Score for pain, Physical activity levels, Additional pain medication, Additional physician/emergency room visits, Sleep, Mood, and Side effects) scores before and after 3 days of treatment. The higher KPS scores(0-100) of patients indicate better quality of life, but the higher SPAASMS scores(0-31) mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jiarong Chen, PhD, Principal Investigator — Affiliated Jiangmen Hospital of Sun Yat-Sen University